CLINICAL TRIAL: NCT01710683
Title: Early Mobilisation Following Discectomy
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled.
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Vejle Hospital (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-07-006
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Reduced Hospital Stay Without Complication
Keywords: Discectomy; 1st postoperative day; Intensive exercise training; Randomized controlled trial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Median age 45 years, 18-63.
  Interventions: Behavioral: Care program
- Intervention group: Median age 46 years, 18-62.
  Interventions: Behavioral: Care program

INTERVENTIONS:
Behavioral: Care program — Care program with multimodal pain treatment including epidural steroid
  Other Names: No other names.
  Groups: Control group
Behavioral: Care program — Care program with multimodal pain treatment including epidural steroid.
  Other Names: No other names.
  Groups: Intervention group

SUMMARY:
After lumbar discectomy 1st postoperative day high intensity exercise training reduced hospital stay, pain and sick leave without side effects in the two year follow-up period.

DETAILED DESCRIPTION:
Postoperative pain is a major cause of delayed convalescence after discectomy. Different analgesic treatments with the use of local analgesics and steroid can reduce the immediate postoperative pain and convalescence after surgery. In orthopaedic and abdominal surgery accelerated stay programs with early mobilisation have reduced pain in the early postoperative periode. The late convalescence after discectomy for herniated disc disease can be reduced with the use of epidural steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary lumbar herniated disc disease who have received and performed a standardized conservative treatment program with intensive exercises.
* Oral and written acceptance.
* Age 18 and above.

Exclusion Criteria:

* Patients with central or lateral spinal stenosis due to spondylosis or disc degeneration who needed bilateral decompression, laminectomy or fusion.
* Patients with cauda equina syndrome who needed acute operative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Northern Orthopaedic Department, Aalborg University Hospital, Denmark; David S. Krum-Moeller, M.D., Study Chair — Department of Orthopaedic Surgery, Vejle and Give Hospital; Lene R. Lauridsen, M.D., Study Chair — Department of Orthopaedic Surgery, Vejle and Give Hospital; Henrik Kehlet, M.D., Study Chair — Section for Surgical Pathophysiology, Juliane Marie Centre, Rigshospitalet, Copenhagen
Locations (1):
- Northern Orthopaedic Division, Aalborg Hospital, Aarhus University, Aalborg, Denmark